CLINICAL TRIAL: NCT02895880
Title: A Risk Assessment Tool to Increase Statin Use Among High Risk Cancer Survivors: Development and Pilot Testing
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1128
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Cancer Survivors; Statin Use Among High Risk Survivors
Keywords: Communication Tool; Cancer Survivors; Increase Statin; 16-1128

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- usual care: first 25 participants will receive usual care (i.e. no risk communication tool)
  Interventions: Behavioral: usual care
- risk communication tool: next 25 participants, clinicians will use the risk communication tool in their discussion about statins and cardiovascular risk reduction
  Interventions: Behavioral: statin communication tool

INTERVENTIONS:
Behavioral: usual care — In order to characterize the content of and variation in usual care, the first 25 patients enrolled in the study will complete a post-visit questionnaire that asks what their doctor told them (if anything) about their risk of cardiovascular disease, risk reduction and statins specifically, and how this information was presented
  Groups: usual care
Behavioral: statin communication tool — The Statin Choice decision aid uses icon arrays to communicate the expected benefits of statins. This modified risk communication tool will maintain the components of the validated original. The adapted paper-based risk communication tool will describe modified risk profiles applicable to the survivors at increased risk for cardiac disease due to chest irradiation.
  Groups: risk communication tool

SUMMARY:
The purpose of this study is to collect initial data on what survivors of childhood, adolescent, and young adult cancer think of how information about statins is communicated. Statins are medications that lower cholesterol. The results of this study will be used to improve the communication about statins. This is to aid patients and their providers in making health care decisions together, also known as shared decision making.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* A personal history of cancer, tumor, or a related illness
* Followed in the Adult Long Term Follow Up Program
* Received ≥ 2000 cGy radiation to the heart/chest
* ≥Ten years post-radiation therapy to the heart/chest
* Age ≥ 25 years old

Exclusion Criteria:

* Evidence of active progression of disease or recurrence
* Neurocognitive deficits that impair ability to give informed consent
* Current use of a statin
* Diagnosis of another primary cancer for which the patient is currently undergoing radiation therapy chemotherapy, or bone marrow transplant
* Diagnosis of CVD with or without current statin use

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Survivorship clinic
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
number of patients who initiated statins after the office visit | 1 year
  This data will allow validation of the adapted tool in the cancer survivor population. Acceptability will be estimated using the tool describe which will be transformed to a 0 to 100 scale and summarized separately in the two populations using means and standard deviations.These preliminary statistics in both populations (intervention and usual care) will be utilized to design a future larger scale study powered to detect a difference between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nirupa Raghunathan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/